CLINICAL TRIAL: NCT06896006
Title: Epidemiological Study of Out-of-hospital Cardiac Arrest in Shenzhen
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-266-01
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-07

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The epidemiology of out-of-hospital cardiac arrest (OHCA) is a significant public health issue, and large-sample studies on such events within China are relatively limited. This study utilizes the Utstein model to evaluate and analyze the epidemiological characteristics of OHCA in Shenzhen from 2011 to 2018. By reviewing ambulance dispatch records and prehospital medical records from the Shenzhen Emergency Medical Center between 2011 and 2018, the study analyzed epidemiological characteristics and reported the results. The main indicators of the study include demographic characteristics such as the gender, age, location of occurrence, key time points, vital signs, chief complaints, and diagnoses of the cases. It also covers prehospital emergency treatment processes, including whether bystanders performed CPR, initial electrocardiogram results, intravenous access establishment, use of epinephrine, defibrillation, tracheal intubation, and other interventions, as well as the outcomes of resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Cases with secondary diagnoses containing only the diagnostic keywords "cardiac arrest" and "sudden death"

Exclusion Criteria:

* 1. Cases with suicide, drowning, advanced cancer, trauma, shock, poisoning, cerebrovascular accidents, etc. 2.Cases with duplicate records for gender, age, time of call, pick-up and drop-off address, and initial diagnosis.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data source consists of ambulance dispatch records and prehospital medical records documented by the Shenzhen Emergency Medical Center from 2011 to 2018.
Sampling Method: Non-Probability Sample
Enrollment: 19672 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Crude incidence rate | 2011-01-01 to 2018-12-31
  The frequency of new cases of a disease in a given population over a given period of time.
Age standardized incidence rate | 2011-01-01 to 2018-12-31
  Incidence rates after removing the influence of age, and incidence rates normalised by age.
Annual percentage change | 2011-01-01 to 2018-12-31
  Indicates the change from one year to the next within a segment at a constant percentage on a log-linear model for evaluating trends within segments.